CLINICAL TRIAL: NCT05357300
Title: Peripheral Nerve Stimulation for Treatment of Chronic Therapy-refractory Sacroiliac Joint Pain
Brief Title: Peripheral Nerve Stimulation for Treatment of Sacroiliac Joint Pain
Acronym: SIlencing
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: PD Dr. med. Simon Bayerl (Other)
Responsible Party: Sponsor-Investigator, PD Dr. med. Simon Bayerl, PD Dr. med., Charite University, Berlin, Germany
Organization: Charite University, Berlin, Germany (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 128236
Record Dates: First submitted 2022-04-26; First posted 2022-05-02 (Actual); Last update posted 2022-05-06 (Actual); Status verified 2022-05

CONDITIONS: Sacroiliac Joint Pain
Keywords: Peripheral Nerve Stimulation; Back Pain; Sacroiliac Joint Pain; Neuromodulation; Persistent Spinal Pain Syndrome
MeSH Terms: conditions — Back Pain

STUDY DESIGN:
Intervention Model Description: Evaluation of the pain reduction in patients treated with peripheral nerve stimulation compared to best medical treatment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peripheral Nerve Stimulation (Active Comparator): Implant of percutaneous leads and impulse generator for peripheral nerve stimulation
  Interventions: Device: Peripheral Nerve Stimulation
- Best Medical Treatment (No Intervention): Physical therapy and therapy with analgetic medication

INTERVENTIONS:
Device: Peripheral Nerve Stimulation — Implant of percutaneous leads for peripheral nerve stimulation of the rami dorsales of the SIJ and gluteal or abdominal implant of impulse generator
  Arms: Peripheral Nerve Stimulation

SUMMARY:
Prospective randomized controlled study, primary objective: Pain reduction in patients with chronic Sacroiliac joint pain after therapy either with Peripheral Nerve Stimulation or with best medical treatment.

Randomization 4:3 to operative (PNS=Peripheral Nerve Stimulation) arm or conservative (BMT= Best Medical Treatment) arm with crossover possibility for the BMT group after 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Subject is at least 18 years old
* Subject with chronic sacroiliac joint pain refractory to conservative treatment
* Subject with NRS of at least 60/100
* Subject with temporary pain reduction of at least 50% (NRS) after fluoroscopy guided SIJ infiltration
* Subject received conservative treatment for at least three months including physiotherapy and pain medication
* Subject is able to understand the study and Impulse generator programming

Exclusion Criteria:

* Pregnancy
* Subject is under age
* Acute traumatic injury of the ISG
* Active inflammation or neoplastic infiltration of the SIJ
* Neoplastic diseases of the spine
* Spinal surgery within the last three months
* The SIJ pain is not the leading symptom
* Contraindication for Neuromodulation Device (severe psychiatric disease, severe coagulation disorder, acute infection, active autoimmune disease with immunosupression)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-04-26 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Change of chronic sacroiliac joint pain | 6 months
  Change of pain measured with a numeric rating scale ranking from minimum 0 to maximum 100 where higher numbers mean a worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Simon H Bayerl, MD, Principal Investigator — Charite University, Berlin, Germany; Dimitri Tkatschenko, MD, Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Charité - Universitätsmedizin Berlin, Department of Neurosurgery, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stinson LW Jr, Roderer GT, Cross NE, Davis BE. Peripheral Subcutaneous Electrostimulation for Control of Intractable Post-operative Inguinal Pain: A Case Report Series. Neuromodulation. 2001 Jul;4(3):99-104. doi: 10.1046/j.1525-1403.2001.00099.x. PMID 22151653
- [Background] van Balken MR, Vandoninck V, Messelink BJ, Vergunst H, Heesakkers JP, Debruyne FM, Bemelmans BL. Percutaneous tibial nerve stimulation as neuromodulative treatment of chronic pelvic pain. Eur Urol. 2003 Feb;43(2):158-63; discussion 163. doi: 10.1016/s0302-2838(02)00552-3. PMID 12565774
- [Background] Al Khalili Y, Jain S, Lam JC, DeCastro A. Brachial Neuritis. 2024 Feb 2. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK499842/ PMID 29763017
- [Derived] Sargut TA, Tkatschenko D, Fruh A, Tuttenberg J, Heckert A, Fleck S, Kuckuck A, Bayerl SH. Study protocol for a prospective, randomized, multicenter trial to investigate the influence of peripheral nerve stimulation on patients with chronic sacroiliac joint syndrome (SILENCING). Trials. 2024 Mar 28;25(1):223. doi: 10.1186/s13063-024-08067-z. PMID 38549128